CLINICAL TRIAL: NCT07104994
Title: Inferior Alveolar Nerve Lateralization and Immediate Dental Implant Placement in Severely Resorbed Mandibles: A Clinical Trial
Brief Title: Inferior Alveolar Nerve Translocation With Dental Implant Placement in Severely Resorbed Mandibles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Science and Technology, Yemen (Other)
Responsible Party: Principal Investigator, Mohammed Ali Al-wesabi, Principal Investigator, University of Science and Technology, Yemen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMFS:14/06/2024
Record Dates: First submitted 2025-07-22; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Sever Mandibular Bone Resorption; Sensory Defect; Implant Failure
Keywords: Inferior Alveolar Nerve; Mandibular Atrophy; Dental Implant; Alveolar Ridge Resorption
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dental implant group (Experimental)
  Interventions: Device: Dental implant

INTERVENTIONS:
Device: Dental implant — insertion of dental implants after surgical tranlocation of the inferior alveolar nerve.

SUMMARY:
This study investigates the effects of inferior alveolar nerve lateralization on the post-implant insertion sensory outcome for patients with severe mandibular bone resorption.

DETAILED DESCRIPTION:
This is a prospective randomized clinical trial. The study was carried out in patients with posterior mandibular atrophies among selected cases from patients attending the Faculty of Dentistry dental polyclinics, and some private dental clinics in Sana'a city The age of patients was above the age of 18 years All patients received a thorough dental examination (extra-oral and intra-oral examination) in dental clinics using a dental mirror, ball-tipped World Health Organization (WHO) dental prob, and dental tweezers. Sterile examination tools by autoclave class B were used. Clinical examination included Oral health and oral hygiene status, interarch distance, dimensions of the edentulous ridge, and soft tissue condition. Panoramic radiographs were taken to assess the condition of the patients' teeth and jawbone, as well as to detect any oral infections requiring treatment. Surgical procedures are performed to translocate the inferior alveolar nerve to provide a good space for implant insertion. All cases ahs undergone follow-up for post-surgical sensory disturbances.

ELIGIBILITY:
Inclusion Criteria:

- All other patients

Exclusion Criteria:

* Patients with active infections, uncontrolled diabetes, history of radiotherapy, chemotherapy, or oral cancer surgery were excluded from this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-04-12 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Cone-beam Computed Tomography (CBCT) | The implant's success rate was determined by primary stability during insertion, assessed by ratchet, and then confirmed by X-ray. CBCTs were taken at 3 months and 4 months after implant insertion to check for marginal bone loss.
  visualize the inferior alveolar canal (IAC) and assess the proximity of the implant to the nerve

SECONDARY OUTCOMES:
Subjective Function Score | Neurosensory evaluation was carried out on the 1st and 7th postoperative day and every month thereafter for up to 6 months.
  Patients rate their perceived sensory function relative to an unaffected area, providing a measure of functional impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Science and technology, Aden, Yemen

REFERENCES:
- [Derived] Hwaiti HS, Al-Rubidi YA, Al-Ashwal A, Al-Hadi Y, Al-Kibsi T, Al-Wesabi MA. Inferior alveolar nerve relocation and immediate dental implant placement in severely resorbed mandibles: a prospective clinical case series. BMC Oral Health. 2025 Dec 13. doi: 10.1186/s12903-025-07492-z. Online ahead of print. PMID 41388273

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT07104994/Prot_SAP_000.pdf